CLINICAL TRIAL: NCT05410327
Title: Historical Trauma and Resilience as a Biological State and Its Association With the Effects of the Traditional Indigenous Food Chokeberry
Brief Title: Health Effects of Traditional Indigenous Chokeberry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Dakota (Other)
Collaborators: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency); Altru Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UND0027177
Record Dates: First submitted 2022-05-26; First posted 2022-06-08 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Inflammation; Mental Health Wellness 1; Oxidative Stress
Keywords: American Indian; Epigenetics; chokeberry; Aronia melanocarpa; Historical Trauma
MeSH Terms: conditions — Inflammation; Historical Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chokeberry consumption (Experimental): Participants will be given 100ml of a water-infused chokeberry juice to consume twice per day for a period of 6 weeks.
  Interventions: Other: Chokeberry (Aronia melanocarpa) juice

INTERVENTIONS:
Other: Chokeberry (Aronia melanocarpa) juice — A water-infused chokeberry (Aronia melanocarpa) juice will be used as the intervention. The brand being used is called 'Superberries'.

SUMMARY:
American Indian populations continue to suffer disproportionately from health problems including such nutrition-related chronic diseases as diabetes and heart disease. This research project will therefore investigate how a traditional Indigenous food called chokeberry (Aronia melanocarpa) impacts epigenetic and metabolic health in relation to resiliency markers in American Indian participants. The process of research with American Indian communities is significant in that it can inform best practices in community engagement orientations, approaches, and models in future research settings.

DETAILED DESCRIPTION:
This study aims to explore the gene expression and metabolic changes that are mediated by consumption of Indigenous chokeberry (Aronia melanocarpa) in adult urban American Indians and to examine the associations between metabolic endpoints, adverse childhood experiences and mental health. The investigators are doing this research study to answer questions about the impact of adult urban American Indians ingesting one of their traditional Indigenous foods called chokeberry on epigenetic, metabolic and mental health markers of trauma and resilience.

For this study, the investigators will be looking to determine:

1. If there are gene expression changes that are mediated by consumption of traditional Indigenous chokeberry in urban adult Great Plains Indians.
2. If there are associations between secondary outcomes such as metabolic endpoints (i.e., 8-OHdG, IL-6, lipids, glucose, CRP, blood pressure), epigenetic states, adverse childhood experiences, and mental health (historical trauma, resiliency, presence of anxiety and depression) in American Indians who have or have not consumed chokeberry as part of a controlled feeding study.

ELIGIBILITY:
Inclusion Criteria:

* Great Plains located American Indians
* Adults between the ages of 18-65

Exclusion Criteria:

* Individuals on blood thinning medications, insulin, those pregnant or breastfeeding and those unable to comply with the research schedule, those who have had stomach or upper gastric resection, those on biologic, chemotherapy and immune suppressant medications, those over 65 years of age due to substantially changing metabolic profiles, and those who have started a new hyperglycemic, hypercholesterolemia, anti-depressant, anti-anxiety, or anti-psychotic medication(s) in the last two months.
* Those who have a current consumption history of chokeberry use (defined by regular use in the last 6 months) or those with a known allergy to chokeberry will also be excluded.
* Those with an acute infection in the last month, those with a vaccination in the last two months, and those on NSAIDS within 93.5 hours of testing may be able to still participate if they do not carry these exclusions in the next testing period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Epigenetics | Baseline and 6 weeks
  The assessment of change in methylation targeted genes

SECONDARY OUTCOMES:
Urinary Hydroxydeoxyguanosine (8-OHdG) | Baseline and 6 weeks
  A commonly used marker of oxidative stress-derived DNA assessed through urine. Assessment of the change in 8-OHdG.
Interleukin 6 (IL-6) | Baseline and 6 weeks
  Is a pro-inflammatory cytokine assessed from the blood that stimulates inflammation. Assessment of the change in IL-6 processes
Lipid panel | Baseline and 6 weeks
  Assessment of the change in HDL, LDL, total cholesterol, triglycerides levels
C-reactive Protein (CRP) | Baseline and 6 weeks
  Measure of systemic inflammation assessed from the blood. Assessment of the change in CRP.
Blood pressure | Baseline and 6 weeks
  Measure of the change in systolic blood pressure and diastolic blood pressure
Patient Health Questionnaire-2 (PHQ-2) | Baseline and 6 weeks
  Validated tool to screen for depression. Assessment of the change PHQ-2 scores. The scale runs from a minimum value of zero to a maximum value of three for each item in the questionnaire. A higher value means a worse outcome.
2-item Generalized Anxiety Disorder Scale (GAD) | Baseline and 6 weeks
  Validated tool to screen for anxiety. Assessment of the change in GAD scores. The scale runs from a minimum value of zero to a maximum value of three for each item in the questionnaire. A higher value means a worse outcome.
Connor-Davidson Resilience Scale 2-item measure (CD-RISC2) | Baseline and 6 weeks
  CD-RISC2 is a brief, self-rated measure of resilience with sound psychometric properties. Assessment of the change in CD-RISC2 scores. Assessment of the change in CD-RISC2 scores. The scale runs from a minimum value of one to a maximum value of four for each item in the questionnaire. A lower value means a worse outcome.
Adverse Childhood Experiences (ACEs) survey (10-item version) | Baseline
  Collects some of the most intensive and frequently occurring sources of stress that children may suffer early in life.
Historical Loss Scale | Baseline
  This scale enumerates perceived losses and asks respondents how frequently these losses came to mind on a 12-item questionnaire specific to Indigenous Peoples. The scale runs from a minimum value of one to a maximum value of six for each item in the questionnaire. A lower value means a worse outcome and is reported in percentage frequency of perceived losses.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Redvers, ND, MPH, Principal Investigator — University of North Dakota School of Medicine & Health Sciences
Locations (1):
- University of North Dakota School of Medicine & Health Sciences, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT05410327/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/27/NCT05410327/ICF_001.pdf